CLINICAL TRIAL: NCT02737982
Title: Sex and Gender Differences in Ischemic Heart Disease: From Bench to Bedside EVA (Endocrine Vascular Disease Approach)
Brief Title: Sex and Gender Differences in Ischemic Heart Disease - Endocrine Vascular Disease Approach
Acronym: EVA
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Ministry of Education, Universities and Research, Italy (Other)
Responsible Party: Principal Investigator, Valeria Raparelli, University Reseacher, University of Roma La Sapienza
Other Study IDs: RBSI14HNVT
Record Dates: First submitted 2016-04-01; First posted 2016-04-14 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Myocardial Ischemia
Keywords: coronary heart disease; gender; platelet; microvascular dysfunction; sexual hormones; cardiac magnetic resonance; percutaneous coronary interventions
MeSH Terms: conditions — Myocardial Ischemia; Coronary Disease; Coitus | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — plasma, serum, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IHD Men: Men with acute or chronic ischemic heart disease undergoing percutaneous coronary interventions
  Interventions: Procedure: percutaneous coronary intervention
- IHD Women: Women with acute or chronic ischemic heart disease undergoing percutaneous coronary interventions
  Interventions: Procedure: percutaneous coronary intervention

INTERVENTIONS:
Procedure: percutaneous coronary intervention — coronary angiography with or without stent implantation, measurement of indexes of epicardial and microvascular reperfusion

SUMMARY:
The application of sex-gender medicine is strongly recommended by World Health Organization and other international organization. In fact, it is emerging that, although men and women are affected to the same cardiovascular diseases (CVD), however they have different risk factors, disease progression and response to pharmacological and not-pharmacological treatments. Consequentially, the identification of biomarkers and therapeutic approaches taking into account sex gender differences (SGD) is relevant to develop a really evidence-based medicine.

With the aim of translate in clinical setting the more recently available basic research evidences on estrogens and androgens balance involvement in modulation of ischemia-reperfusion myocardial damage, the investigators planned to conduct a research study on patients, affected by suspected or known ischemic heart disease (IHD) undergoing angiography and/or percutaneous coronary interventions (PCI), aged more than 18 years of both sex in ratio 1:1. Thus, in this setting, the goals of this proposal are:

1. To assess the sex-gender difference in entity of microvascular reperfusion damage in patients with IHD undergoing urgent or elective PCI;
2. To evaluate estrogen/androgen-dependent and -independent effects in gender-related differences on myocardial ischemia reperfusion damage occurring during PCI;
3. To investigate the differences in terms of platelet biology between men and women affected by IHD undergoing urgent or elective PCI, matched for age and clinical cardiovascular and metabolic characteristics;
4. To verify sex-driven interplay between response to PCI procedure, platelet function, sex hormones and entity of reperfusion and myocardial damage, as well as, the impact on clinical outcomes during a 1-year follow up.

This research study wants to explore and consequently elucidate biological mechanisms responsible for sex-based differences in vivo human models of ischemia reperfusion myocardial damage. Moreover, the investigators expected to clarify the impact of biological variables evaluated on clinical outcomes after reperfusion therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients with ischemic heart disease (acute or chronic) undergoing percutaneous coronary intervention (urgent or elective)
* written informed consent
* both sex
* aged more than 18 years

Exclusion Criteria:

* patients with expectancy of life less than 12 months
* active cancer
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women who referred with a suspected IHD to the cath-lab for undergoing percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Assessment of corrected Thrombolysis In Myocardial Infarction frame count and myocardial blush grade | baseline; within 1h from PCI
  angiographic assessment of coronary flow

SECONDARY OUTCOMES:
Sexual hormones levels in patients with IHD undergoing PCI | baseline
  Evaluation and impact of sexual hormones levels in gender-related differences during myocardial reperfusion
Platelet activation markers including Thromboxane, soluble cluster designation 40 (CD40) Ligand and soluble P-selectin in patients with IHD undergoing PCI | baseline; within 1h from PCI; 12 months
  Evaluation of Sex and gender differences in platelet function
Clinical outcomes including cardiovascular mortality, re-hospitalization and restenosis | 12 months
Microvascular dysfunction assessed by cardiac magnetic resonance | 7 days from percutaneous coronary intervention
  Among the EVA registry, we plan to perform a pilot study including: patients with stable angina with mono-vessel obstructive coronary artery disease (CAD) undergoing PCI; patients with stable angina undergoing angiography that documented no obstructive coronary disease (with a stenosis <50%) with a impairment of microvascular dysfunction defined during angiography by a myocardial blush grade <2 or coronary flow reserve <2 after stress stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Raparelli, MD, Principal Investigator — Experimental Medicine Department, Sapienza University of Rome
Locations (1):
- Policlinico Umberto I , Sapienza University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Raparelli V, Romiti GF, Di Teodoro G, Seccia R, Tanzilli G, Viceconte N, Marrapodi R, Flego D, Corica B, Cangemi R, Pilote L, Basili S, Proietti M, Palagi L, Stefanini L; EVA Investigators. A machine-learning based bio-psycho-social model for the prediction of non-obstructive and obstructive coronary artery disease. Clin Res Cardiol. 2023 Sep;112(9):1263-1277. doi: 10.1007/s00392-023-02193-5. Epub 2023 Apr 1. PMID 37004526
- [Derived] Raparelli V, Proietti M, Romiti GF, Lenzi A, Basili S; EVA Collaborative Group. The Sex-Specific Detrimental Effect of Diabetes and Gender-Related Factors on Pre-admission Medication Adherence Among Patients Hospitalized for Ischemic Heart Disease: Insights From EVA Study. Front Endocrinol (Lausanne). 2019 Feb 25;10:107. doi: 10.3389/fendo.2019.00107. eCollection 2019. PMID 30858826
- [Derived] Raparelli V, Proietti M, Lenzi A, Basili S; EVA Collaborators. Sex and Gender Differences in Ischemic Heart Disease: Endocrine Vascular Disease Approach (EVA) Study Design. J Cardiovasc Transl Res. 2020 Feb;13(1):14-25. doi: 10.1007/s12265-018-9846-5. Epub 2018 Dec 3. PMID 30511337